CLINICAL TRIAL: NCT06076655
Title: The Effectiveness of Exercise and Mobilization in Correcting Deformity in Children With Diplegic Cerebral Palsy With Hallux Valgus
Brief Title: Hallux Valgus Treatment Developed for Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Bedia ÖZDEMİR, Physiotherapist, Istanbul Arel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulArelUBediaozdemir
Record Dates: First submitted 2023-10-01; First posted 2023-10-11 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Hallux Valgus
Keywords: HALLUX VALGUS; CEREBRAL PALSY; EXERCISE; MOBILIZATION
MeSH Terms: conditions — Hallux Valgus; Cerebral Palsy; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EXERCISE AND MOBILIZATION PROGRAM — EXERCISE AND MOBILIZATION PROGRAM The Hallux Valgus exercise program determined by the physiotherapist will be applied twice a week in the rehabilitation unit under the supervision of a physiotherapist. Each exercise and mobilization will be planned as 2 sets of 10 repetitions and 15 seconds between sets, and will be carried out throughout the interval for 12 weeks. In addition, home exercises will be given twice a day, and each exercise will be followed in 2 sets of 10 repetitions with a 15-second interval between sets.
  The exercise and mobilization program planned to be implemented in this study for children with diplegic cerebral palsy is an exercise and mobilization program that has yielded positive results in various studies in adults. We created a sample protocol with exercise and mobilization practices that were found effective in these studies.

SUMMARY:
This study is a clinical trial.Hallux valgus, one of the common deformities in the foot in children with diplegic Cerebral Palsy, has caused serious problems in daily life activities in children and has usually resulted in surgical operation. Due to the lack of sufficient studies on this topic, our aim in our study is to show the importance of exercise and mobilization applied by physiotherapists in the early stages of hallux valgus deformity, which is common in children with Cerebral palsy, in correcting the deformity, and an example exercise program for physiotherapists.

The study will include 15 individuals with cerebral palsy diagnosed with hallux valgus by a physician at the Physiotherapy and Rehabilitation clinic at Istanbul FSM Madenler Medical Center according to the following criteria. Children diagnosed with diplegic SP, aged 9-16, with Communication Function Classification System Levels 1 and 2, ambulation level GMFCS 1-2, using AF Dec and GRAPHO and without any auxiliary device use, Manchester scale stages 1 and 2 will be included. Those who cannot walk independently, GMSCS 3 and above, children using assistive devices, Communication Function Classification System Level 3 and above, children with Manchester scale Stage 3 hallux valgus will be excluded from the study.Manchester November Scale for Hallux valgus classification, Hallux valgus angle and Foot and Ankle joint range of motion goniometer, Spasticity Modified Ashworth Scale (MAS), Foot and Ankle muscle strength Kendall Manual Muscle Strength Assessment, Pain Visual Analogue Scale (VAS), Communication skill Communication Function Classification System with Gross Motor Function Classification System GMFCS level, American orthopedic foot-ankle association-hallux MTF-IF scale evaluation is planned.

DETAILED DESCRIPTION:
EXERCISE PROGRAM The Hallux Valgus exercise program determined by the physiotherapist will be performed twice a week in the rehabilitation unit accompanied by a physiotherapist, each exercise and mobilization will be planned as 2 sets of 10 repetitions and 15 seconds between sets, and will be performed for 12 weeks Dec. In addition, home exercises will be given 2 times a day and each exercise will be followed by 10 repetitions for 2 sets and 15 seconds Dec between sets.

The exercise and mobilization program planned to be implemented in this study for children with diplegic Cerebral Palsy is an exercise and mobilization program that has shown positive results in adults in various studies. We have created an exemplary protocol with the exercise and mobilization practices that were found effective in these studies. Below is our sample program.

Exercise and mobilization program to be implemented in the clinic accompanied by a physiotherapist:

1. 1. Metatarsophalangeal Joint (MTFE) mobilization

   * 1. MTF Traction mobilization
   * 1. MTF medial and lateral shift mobilization
   * 1. MTF dorso-plantar mobilization
   * 1. MTF sesamoid mobilization
2. Passive thumb abduction with thumb traction from the first metatarsophalangeal joint
3. Toe Sequential Exercises

   * 1. Phase: Bringing all the fingers into extension without breaking the contact of the heel and metatarsal heads with the ground.
   * 2. Phase: While the other fingers are still in extension, the smallest finger is moved laterally and flexibly to make contact with the ground again.
   * 3. Phase: Ensuring contact with the ground by slowly and controllably bringing the thumb into abduction and flexion while the other fingers maintain the position they took last
4. Active thumb abduction
5. Thumb abduction exercise with toe toe exercise rubber
6. The movement of collecting sheets for active flexion of the ind November muscles of the foot
7. Ball rolling exercise on the sole of the foot
8. Active stretching exercise of the gastro-soleus November
9. Hamstring November muscle active stretching exercise (Rose et al., 2020; Okur et al., 2019; Kim M-H et al.,2015)

Home exercise program to be given to the patient:

1. Toe Sequential Exercises

   * 1. Phase: Bringing all the fingers into extension without breaking the contact of the heel and metatarsal heads with the ground.
   * 2. Phase: While the other fingers are still in extension, the smallest finger is moved laterally and flexibly to make contact with the ground again.
   * 3. Phase: Ensuring contact with the ground by slowly and controllably bringing the thumb into abduction and flexion while the other fingers maintain the position they took last
2. Active thumb abduction
3. Thumb abduction exercise with Toe Toe Exercise Rubber
4. The movement of collecting sheets for active flexion of the ind November muscles of the foot
5. Ball rolling exercise on the sole of the foot
6. Active stretching exercise of the gastro-soleus November
7. Hamstring November muscle active stretching exercise

Evaluations will be performed 3 times before treatment, in the middle of treatment and at the end of treatment.

Exercise and mobilization performed alone as a result of treatment will prevent hallux valgus of seals in children with diplegic cerebral palsy, prevent surgical operation and provide an exemplary exercise protocol to physiotherapists.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with cerebral palsy,
* Being a spastic diplegic type of cerebral palsy,
* Age range 9-16,
* Communication Function Classification System Level 1 and 2,
* Children with ambulatory level GMFCS 1-2,
* Using AFO and GRAFO,
* Children who do not use any assistive devices,
* Children with Manchester scale Stage 1 and 2 hallux valgus will be included in the study.

Exclusion Criteria:

* Those who cannot walk independently,
* GMSCS 3 and above,
* Does not use AFO and GRAFO,
* Children using assistive devices,
* Communication Function Classification System Level 3 and above,
* Manchester scale stage 3 hallux valgus,
* Children with spasticity values above 1+ according to the Modified Ashworth Scale will be excluded from the study.

Ages: 117 Months to 201 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-10-02 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
COMMUNICATION FUNCTION CLASSIFICATION SYSTEM (CFCS) | ONLY BEFORE TREATMENT
  The aim of the communication function classification system is to classify daily communication performance between I and V levels in individuals with Cerebral Palsy.Dec.This classification is carried out with a form.Our aim is to include individuals who can express themselves in our study. Level 1 represents the effective receiver and transmitter with familiar and foreign partners, level 5 rarely represents the effective transmitter and receiver, even with familiar partners.
GROSS MOTOR FUNCTİON CLASSİFİCATİON SYSTEM | ONLY BEFORE TREATMENT
  Gross motor function in children with cerebral palsy is a standardized method that classifies motor function differences, especially in sitting and walking, into 5 levels. Level I walks without restriction; Level II walks with restrictions; Level III walks using hand-held mobility devices; Level IV, independent self-mobility limited and may use motorized mobility device; Level V is transported in a hand-propelled wheelchair.
USE OF ORTHOSES AND ASSISTIVE DEVICES | ONLY BEFORE TREATMENT
  A crıterıa has been prepared to questıon ıf there ıs an orthosıs ın the lower extremıtıty that chıldren wıth cerebral palsy use ın daıly lıfe, ıf any, what type of orthoses ıt ıs, and ıf they use assıstıve devıces.
PARTICIPANT EVALUATION FORM | ONLY BEFORE TREATMENT
  The sociodemographic characteristics of the children were recorded and information such as name, surname, age, height, weight, gender, and body mass index were questioned. Factors causing the disease, accompanying diseases and extremity involvement are determined and recorded in the evaluation form.

SECONDARY OUTCOMES:
MANCHESTER SCALE | BEFORE TREATMENT ,MIDDLE OF TREATMENT, AT THE END OF TREATMENT
  This scale, which was developed to determine the degree of hallux valgus deformity in individuals; It is considered at 4 levels: none (1), mild (2), moderate (3), and severe (4) and is used as a clinical tool that includes photographs of the foot.Measurements were made 3 times before starting treatment, in the middle of treatment and at the end of treatment.
HALLUX VALGUS ANGLE | BEFORE TREATMENT ,MIDDLE OF TREATMENT, AT THE END OF TREATMENT
  Measurements will be made using a universal goniometer. The first metatarsophalangeal joint was determined as the pivot point, and one arm of the goniometer was placed parallel to the articular joint. The first metatarsal bone is parallel to the proximal phalanx of the other arm and the hallux angle is recorded in degrees. Individuals with a toe hallux angle over 15 degrees are considered to have Hallux valgus. Measurements were taken 3 times before starting treatment, in the middle of treatment and at the end of treatment.
KENDALL MANUAL MUSCLE STRENGTH ASSESSMENT | BEFORE TREATMENT ,MIDDLE OF TREATMENT, AT THE END OF TREATMENT
  It will be used to evaluate November's muscle strength in children. This Test is scored Decently between 0 and 5.0 is the worst, 5 gives the best value. November November, the muscle groups to be evaluated were; MTF Flexion and Extension, IF Flexion and IF Extension Abduction of the big toe, plantar flexion of the ankle, dorsiflexion, eversion and inversion muscle groups were applied. Each assessment was repeated three times and the average was taken.
VİSUAL ANALOGUE SCALE | BEFORE TREATMENT ,MIDDLE OF TREATMENT, AT THE END OF TREATMENT
  It is used to evaluate possible change in pain intensity. It will be reported as no pain (0) and the worst pain imaginable (10). And the subjects will be asked to mark their pain at rest. Then, the marks on this line will be measured in centimeters and the results will be recorded. Measurements were taken 3 times before starting treatment, in the middle of treatment and at the end of treatment.
AMERICAN ORTHOPEDIC FOOT-ANKLE ASSOCIATION HALLUX INTERPHALANGEAL JOINT SCALE | BEFORE TREATMENT ,MIDDLE OF TREATMENT, AT THE END OF TREATMENT
  This 100-point scale is used to evaluate subjective and objective factors. Pain is evaluated as 40 points; function is evaluated as 45 points and alignment is evaluated as 15 points for a total of 100 points. If the patient has bilateral deformity, the result characteristics indicating the foot problem are recorded separately for both feet.Measurements were made 3 times before starting treatment, in the middle of treatment and at the end of treatment.
MODIFIED ASHWORTH SCALE | BEFORE TREATMENT ,MIDDLE OF TREATMENT, AT THE END OF TREATMENT
  Modified Ashworth Scale (MAS) is used for spasticity. Hip Flexors, Hip Adductors, Rectus Femoris and hamstring muscle groups, Foot-ankle plantar flexion and dorsiflexion will be evaluated while the children lie on their backs in a comfortable position in bed. MAS is a 6-point scale that evaluates muscle tone.
  0: No increase in tone and 4: Indicates that the involved part is rigid in flexion or extension. Measurements were made 3 times before starting treatment, in the middle of treatment and at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: BEDİA ÖZDEMİR, Principal Investigator — Istanbul Arel University; SEÇİL ÖZKURT, Study Chair — Istanbul Arel University; OLCAY GÜLER, Study Chair — Istanbul Arel University

IPD SHARING:
Plan to Share IPD: Yes
It is planned that our individual participant data will be shared by mail with people who meet the appropriate Access Criteria.
Supporting Information: Study Protocol
Time Frame: Dec January October 2023 to January 2024 is planned for our study.
Access Criteria: * Magazine editor
  * Members of the ethics committee

REFERENCES:
- [Background] Kim MH, Yi CH, Weon JH, Cynn HS, Jung DY, Kwon OY. Effect of toe-spread-out exercise on hallux valgus angle and cross-sectional area of abductor hallucis muscle in subjects with hallux valgus. J Phys Ther Sci. 2015 Apr;27(4):1019-22. doi: 10.1589/jpts.27.1019. Epub 2015 Apr 30. PMID 25995546
- See also: The effects of taping and foot exercises on patients with hallux valgus: a preliminary study — https://doi.org/10.3906/sag-0912-499
- See also: EVALUATION OF THE EFFICACY OF MANUAL MOBILIZATION TECHNIQUES IN THE TREATMENT OF HALLUX RIGIDUS: CASE SERIES — https://dergipark.org.tr/tr/download/article-file/642859